CLINICAL TRIAL: NCT04639245
Title: ATTAMAGE-A1.: Phase I/II Study of Autologous CD8+ and CD4+ Transgenic T Cells Expressing High Affinity MAGE-A1-Specific T-Cell Receptor (TCR) Combined With Atezolizumab in Patients With Metastatic MAGE-A1 Expressing Cancer
Brief Title: Genetically Engineered Cells (MAGE-A1-specific T Cell Receptor-transduced Autologous T-cells) and Atezolizumab for the Treatment of Metastatic Triple Negative Breast Cancer, Urothelial Cancer, or Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: SignalOne Bio, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Schweizer, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1007463; NCI-2020-06602 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10420 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-11-13; First posted 2020-11-20 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Triple-Negative Breast Carcinoma; Metastatic Urothelial Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Triple Negative Breast Neoplasms; Carcinoma, Transitional Cell; Lung Neoplasms | interventions — atezolizumab; Cyclophosphamide; fludarabine; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (FH-MagIC TCR-T cells, atezolizumab) (Experimental): LYMPHODEPLETION: Patients receive cyclophosphamide IV and fludarabine IV on days -4, -3, and -2 before each T-cell infusion.
  T-CELL INFUSION: Patients receive FH-MagIC TCR-T cells IV over 15-20 minutes. Six to twelve weeks after first T-cell infusion, patients with progressive disease and non-persisting transgenic TCR T cells may receive a second T-cell infusion.
  In the Phase 2 portion of the study, atezolizumab will be administered as standard of care beginning 24-72 hours after T-cell infusion. Atezolizumab will be given IV every 3 weeks for at least 1 year in the absence of disease progression or unacceptable toxicity. An alternative PD1 inhibitor may be substituted if atezolizumab (preferred) is not available.
  Interventions: Drug: Atezolizumab; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: MAGE-A1-specific T Cell Receptor-transduced Autologous T-cells; Biological: PD1 Inhibitor

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Biological: MAGE-A1-specific T Cell Receptor-transduced Autologous T-cells — Given IV
  Other Names: MAGE-A1-specific T Cell Receptor-transduced Autologous CD8+ and CD4+ T-cells; MAGE-A1-specific TCR-transduced Autologous T-cells
Biological: PD1 Inhibitor — Given IV
  Other Names: PD-1 Inhibitor; PD-1-targeting Agent; Programmed Cell Death Protein 1 Inhibitor; Protein PD-1 Inhibitor; Anti-PD-1 Agent

SUMMARY:
This phase I/II trial investigates the side effects of genetically engineered cells called FH-MagIC TCR-T cells and how well they work with atezolizumab in treating patients with triple negative breast cancer, urothelial cancer, or non-small cell lung cancer that has spread to other places in the body (metastatic). T cells are infection fighting blood cells that can kill tumor cells. The T cells given in this study will come from the patient and will have a new gene put in them that makes them able to recognize MAGE-A1, a protein on the surface of tumor cells. These MAGE-A1-specific T cells may help the body's immune system identify and kill MAGE-A1 tumor cells. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving FH-MagIC TCR-T cells with atezolizumab may help treat patients with triple negative breast cancer, urothelial cancer, or non-small cell lung cancer.

DETAILED DESCRIPTION:
OUTLINE:

This is a phase I, dose escalation study of FH-MagIC TCR-T cells followed by a phase II study.

LYMPHODEPLETION: Patients receive cyclophosphamide intravenously (IV) and fludarabine IV on days -4, -3, and -2 before each T-cell infusion.

T-CELL INFUSION: Patients receive FH-MagIC TCR-T cells IV over 15-20 minutes. Six to twelve weeks after first T-cell infusion, patients with progressive disease and non-persisting transgenic TCR T cells may receive a second T-cell infusion.

In the Phase 2 portion of the study, atezolizumab will be administered as standard of care beginning 24-72 hours after T-cell infusion. Atezolizumab will be given IV every 3 weeks for at least 1 year in the absence of disease progression or unacceptable toxicity. An alternative PD1 inhibitor may be substituted if atezolizumab (preferred) is not available.

After completion of study treatment, patients are followed up annually for 15 years after final infusion of FH-MagIC TCR-T.

ELIGIBILITY:
Inclusion Criteria:

* Tissue confirmation of triple negative breast cancer (TNBC), urothelial carcinoma or non-small cell lung cancer (NSCLC) and expression of MAGEA1: Participants must have metastatic disease. Confirmation of diagnosis must be or have been performed by internal pathology review of archival, initial or subsequent biopsy or other pathologic material at Fred Hutchinson Cancer Research Center (FHCRC)/Seattle Cancer Care Alliance (SCCA)/University of Washington Medical Center (UWMC). Patients with TNBC must meet the American Society of Clinical Oncology - College of American Pathologists (ASCO-CAP) definition of negative estrogen, progesterone and HER2 receptor expression. Baseline tissue will be stained to confirm MAGE-A1 expression
* Measurable disease by RECIST 1.1 criteria: Participants must have measurable disease, defined as at least one target lesion that can be measured in at least one dimension (longest diameter to be recorded) as >= 10 mm, unless lymph node in which case short axis must be >= 15 mm. Baseline imaging (for example diagnostic computed tomography [CT] chest/abdomen/pelvis and imaging of the affected extremity as appropriate), brain imaging (magnetic resonance imaging [MRI] or CT scan) must be obtained within 45 days of prior to start of first planned FH-MAGEA1-A2TCR infusion. MRI can be substituted for CT in patients unable to have CT contrast. Measurable disease is not required for purposes of leukapheresis /cell manufacturing storage for patients who meet HLA and expression criteria but not standard treatment criteria
* Previous treatment with standard of care (SOC) Food and Drug Administration (FDA)-approved therapies. Patients with NSCLC who have actionable somatic mutations or alterations in EGFR, ROS1 and ALK with FDA-approved drug therapy options will be eligible for study only after treatment with targeted therapies for those mutations have been offered or received. Patients with urothelial carcinoma who are candidates for enfortumab vedotin (enfortumab vedotin-ejfv) will be eligible for study after prior treatment with enfortumab vedotin-ejfv has been offered or received

  * Note: Participants will be eligible to enroll before standard therapy is received in order to expedite leukapheresis/cell manufacturing as long as the aforementioned agent is administered prior to lymphodepletion and/or cell infusion
* Previous treatment with PD-1 axis inhibitor: Patients in Phase I/2 must have been offered or been previously treated with at least one dose of a PD-L1 axis inhibitor (e.g. PD-1 or PD-L1 inhibiting monoclonal antibody such as pembrolizumab, nivolumab, avelumab, atezolizumab, durvalumab). If received, they must have either developed progression or still have detectable disease and not have developed Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher toxicity while on treatment. Patients may have received 1 or more prior systemic regimens for metastatic TNBC or NSCLC. There is no upper limit on prior regimens. Patients may have received prior anti-PD-1/anti-PD-L1 in the neoadjuvant or adjuvant setting
* HLA type HLA-A*02:01: Participants must be HLA-A*02:01 in order for infused transgenic T cells in order to insure recognition of antigen-MHC complexes. HLA typing should be determined though a molecular approach in a clinical laboratory licensed for HLA typing
* Life expectancy must be anticipated to be > 3 months at trial entry
* 18 years or older
* Capable of understanding and providing a written informed consent
* If fertile, willingness to comply with reproductive requirements
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Tumor tissue amenable to safe biopsy and subject willing to undergo serial tumor biopsies: Should there be no tumor tissue that is accessible for biopsy, patients will still be considered for participation, at discretion of the sponsor and in consultation with the investigator. Similarly, should an investigator determine that a biopsy cannot be performed safely for clinical reasons biopsies may be cancelled or retimed after confirming plan with the sponsor
* Participants must be at least three weeks from last systemic treatment at the time of cell collection: At least 3 weeks must have passed since any: immunotherapy (for example, T-cell infusions, immunomodulatory agents, interleukins, vaccines), small molecule or chemotherapy cancer treatment, other investigational agents. There is no washout period for radiation, so long as radiated lesion is not the lesion being evaluated for RECIST measurements on the protocol. Bisphosphonates are permitted but the concurrent treatment with RANK ligand inhibitors (i.e., denosumab) is not permitted within 8 weeks of treatment
* Serum creatine < 2.5 mg/dL or estimated glomerular filtration rate (eGFR) > 30 mL/min
* Total bilirubin (tBili) < 3.0 mg/dL. Patients with suspected Gilbert syndrome may be included if Tbili > 3 but no other evidence of hepatic dysfunction
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 x upper limit of normal (ULN)
* =< grade 1 dyspnea and oxygen saturation (SaO2) >= 92% on ambient air. If pulmonary function tests (PFTs) are performed based on the clinical judgement of the treating physician, patients with forced expiratory volume in 1 second (FEVI) >= 50% of predicted and carbon monoxide diffusing capability test (DLCO) (corrected) of >= 40% of predicted will be eligible
* Patients 60 years of age or older are required to have left ventricular ejection fraction (LVEF) evaluation performed within 60 days prior to enrollment. LVEF may be established with echocardiogram or multigated acquisition scan (MUGA) scan, and left ejection fraction must be >= 35%. Cardiac evaluation for other patients is at the discretion of the treating physician
* Absolute neutrophil count (ANC) > 500 cells/ mm^3

Exclusion Criteria:

* Expression of HLA B*4901: participants will be excluded due to the risk of alloreactivity
* Participants of childbearing potential must have a negative serum pregnancy test within 14 days prior to enrollment. Childbearing potential is defined as women who have not been surgically sterilized and who are not postmenopausal (free of menses for at least 1 year)
* Patients with active autoimmune disease requiring immunosuppressive therapy are excluded. Case-by-case exemptions are possible with approval by principal investigator (PI)
* Prior solid organ transplant or allogenic hematopoietic stem cell transplant: Kidney transplant patients will be considered on a case-by-case basis requiring discussion with PI. If kidney transplant, patient must have dialysis access, dialysis plan, supportive nephrologist, willingness to stop transplant immunosuppression, and express understanding that rejection is possible outcome. Dialysis or costs related to transplant kidney will not be supported by the study. Participants having had any other solid organ transplants will be excluded, as will those with any history of allogeneic stem cell transplant
* Corticosteroid therapy at a dose equivalent of > 0.5 mg/kg of prednisone-equivalent per day
* Concurrent use of other investigational anti-cancer agents
* Chronic lymphocytic leukemia (CLL) or other active hematologic malignancy
* Active uncontrolled infection: Human immunodeficiency virus (HIV) positive participants on highly active anti-retroviral therapy (HAART) with a CD4 count > 500 cells/mm^3 are considered controlled, as are individuals with a history of hepatitis C who have successfully completed antiviral therapy with an undetectable viral load, and those with hepatitis B who have, per standard practice, hepatitis well-controlled on medication (e.g., AST and ALT < 5 x ULN)
* Participants may not have uncontrolled or concurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Participants with small asymptomatic brain metastases (< 1 cm) or those with brain metastases previously treated with surgery or radiotherapy will be considered for inclusion at discretion of principal investigator, so long as other eligibility criteria are met.
* For patients in phase 1/2, grade 3 or higher immune-mediated toxicity to any prior PD-L1 axis blocking agent
* Active treatment for prior immune related adverse event to any immunotherapy: Participants receiving ongoing treatment for prior serious immune related adverse events are excluded, with exception of hormone supplementation or corticosteroid therapy at equivalent of up to 0.5 mg/kg prednisone per day, unless otherwise approved by PI
* Study participants must not have significant active underlying neurologic disease, unless approved by PI. Neuropathy related to diabetes or prior chemotherapy is acceptable
* Other medical, social, or psychiatric factor that interferes with medical appropriateness and/or ability to comply with study, as determined by the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schweizer, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wermke M, Holderried TAW, Luke JJ, Morris VK, Alsdorf WH, Wetzko K, Andersson BS, Wistuba II, Parra ER, Hossain MB, Grund-Groschke S, Aslan K, Satelli A, Marisetty A, Satam S, Kalra M, Hukelmann J, Kursunel MA, Pozo K, Acs A, Backert L, Baumeister M, Bunk S, Wagner C, Schoor O, Mohamed AS, Mayer-Mokler A, Hilf N, Krishna D, Walter S, Tsimberidou AM, Britten CM. First-in-human dose escalation trial to evaluate the clinical safety and efficacy of an anti-MAGEA1 autologous TCR-transgenic T cell therapy in relapsed and refractory solid tumors. J Immunother Cancer. 2024 Jul 22;12(7):e008668. doi: 10.1136/jitc-2023-008668. PMID 39038917

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (FH-MagIC TCR-T Cells, Atezolizumab): LYMPHODEPLETION: Patients receive cyclophosphamide IV and fludarabine IV on days -4, -3, and -2 before each T-cell infusion.
  T-CELL INFUSION: Patients receive FH-MagIC TCR-T cells IV over 15-20 minutes. Six to twelve weeks after first T-cell infusion, patients with progressive disease and non-persisting transgenic TCR T cells may receive a second T-cell infusion.
  In the Phase 2 portion of the study, atezolizumab will be administered as standard of care beginning 24-72 hours after T-cell infusion. Atezolizumab will be given IV every 3 weeks for at least 1 year in the absence of disease progression or unacceptable toxicity. An alternative PD1 inhibitor may be substituted if atezolizumab (preferred) is not available.
  Atezolizumab: Given IV
  Cyclophosphamide: Given IV
  Fludarabine: Given IV
  MAGE-A1-specific T Cell Receptor-transduced Autologous T-cells: Given IV
  PD1 Inhibitor: Given IV
Period: Overall Study
Arm/Group | Treatment (FH-MagIC TCR-T Cells, Atezolizumab)
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (FH-MagIC TCR-T Cells, Atezolizumab)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants That Experienced Treatment-related Unexpected Grade 3 or Higher Adverse Events
Time Frame: 4 weeks post last infusion per patient
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (FH-MagIC TCR-T Cells, Atezolizumab)
Number analyzed (Participants) | 1
Participants | 0

2. Primary Outcome: Best Overall Response
Description: Lesions will be separately tracked but response determined in totality. As indicated, patient must have at least one trackable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Response will be a defined as best overall response by RECIST 1.1. A Complete Response will be defined as total regression of all tumors, a Partial Response as 30% or greater decrease in the sum of the longest diameter of target lesions compared to baseline and Progressive Disease as 20% increase in the sum of the longest diameter of target lesions compared to the smallest prior diameter. If the disease does not fall in either category it will be considered Stable Disease (RECIST v1.1 criteria).
Time Frame: 1 year post infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (FH-MagIC TCR-T Cells, Atezolizumab)
Number analyzed (Participants) | 1
Participants
  Complete response | 0
  Partial response | 0
  Stable disease | 1
  Progressive disease | 0

3. Secondary Outcome: Peripheral Blood Concentration of Infused Transgenic T Cells Over Time
Description: Results will be reported by sample for the single treated patient. Patient samples were tested using a WPRE assay showing transgenic T cells in blood. This was detected by qPCR.
Time Frame: 1 year post infusion
Measure: Number; unit: WPRE copies/Cell
Arm/Group | Treatment (FH-MagIC TCR-T Cells, Atezolizumab)
Number analyzed (Participants) | 1
WPRE copies/Cell
  BU712PRETX | 0.0
  BU712I1D000 | 0.0
  BU712I1D001 | 0.0101
  BU712I1D003 | 0.0303
  BU712I1D007 | 0.0379
  BU712I1D014 | 0.0379
  BU712I1D021 | 0.0111
  BU712I1D028 | 0.0087
  BU712I1D056 | 0.0107
  BU712I1D180 | 0.0062
  BU712I2D03 | 0.1167
  BU712I2D07 | 0.0795
  BU712I2D14 | 0.0353
  BU712I2D21 | 0.0267
  BU712I2D28 | 0.0333
  BU712I2D56 | 0.0027
  BU712I2D84 | 0.0070

4. Secondary Outcome: Participants That Displayed Transgenic T Cells in Tumor Tissue
Description: Outcome will be reported as a count of participants that displayed transgenic T cells in their tumor tissue after treatment. This was assessed by WRPE staining and scRNA sequencing. Unfortunately, no transgenic cells were detected on the one treated patient's tumors.
Time Frame: 1 year post infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (FH-MagIC TCR-T Cells, Atezolizumab)
Number analyzed (Participants) | 1
Participants | 0

5. Secondary Outcome: Progression-free Survival
Description: Outcome will be reported as a count of participants that were alive as the 1 year post infusion timepoint and also had not experienced progression at that timepoint.
Time Frame: 1 year post infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (FH-MagIC TCR-T Cells, Atezolizumab)
Number analyzed (Participants) | 1
Participants | 0

6. Secondary Outcome: Overall Survival
Description: Outcome will be reported as a count of participants that were alive at the 1 year post infusion timepoint.
Time Frame: 1 year post infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (FH-MagIC TCR-T Cells, Atezolizumab)
Number analyzed (Participants) | 1
Participants | 0

7. Secondary Outcome: Objective Response Rates
Description: Evaluated by immune-related RECIST criteria. Outcome will be reported as a count of participants that experienced a Complete Response or Partial Response per RECIST criteria. A complete response (CR) will be defined as total regression of all tumors, a Partial Response as 30% or greater decrease in the sum of the longest diameter of target lesions compared to baseline and Progressive Disease as 20% increase in the sum of the longest diameter of target lesions compared to the smallest prior diameter. If the disease does not fall in either category it will be considered Stable Disease (RECIST v1.1 criteria).
Time Frame: 1 year post infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (FH-MagIC TCR-T Cells, Atezolizumab)
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 4 weeks following the last infusion per patient.
Arm/Group | Treatment (FH-MagIC TCR-T Cells, Atezolizumab)
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (FH-MagIC TCR-T Cells, Atezolizumab) (N=1)
Bloating (Gastrointestinal disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Dizziness (Nervous system disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Hyperphosphatemia (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (3)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: First half of document: pages 1-40 (File size too large) (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT04639245/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: Second half of document: pages 41-78 (File size too large) (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT04639245/Prot_SAP_002.pdf
  • Informed Consent Form (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04639245/ICF_000.pdf